CLINICAL TRIAL: NCT06407076
Title: Strengths and Weaknesses of Physiotherapy in the Daily Work of an Intensive Care Unit: A Qualitative Study
Brief Title: Strengths and Weaknesses of Physiotherapy in the Daily Work of an Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: University of Oviedo (Other)
Responsible Party: Principal Investigator, Ruben Cuesta Barriuso, Principal Investigator, University of Oviedo
Other Study IDs: FisUCI
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-05

CONDITIONS: Healthcare
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observacional group: 18 people (6 doctors, 6 nurses and 6 physiotherapists) will be included in the study. The 18 health professionals will participate in personal interviews and focus groups (3 focus groups with 6 participants each). Participants will be recruited from the Intensive Care Unit of the Hospital Universitario Central de Asturias.
  Interventions: Other: Interviews

INTERVENTIONS:
Other: Interviews — Following the design of the questionnaire, using open-ended questions based on the availability, accessibility, acceptability and quality (AAAQ) framework, qualitative semi-structured personal interviews were used to collect the data. In this way it was possible to collect information in a more detailed way. The subjects included in the study had to answer the questions posed by the main researcher, responding with open or closed answers, through a questionnaire created for this purpose.

SUMMARY:
Background. A stay in the Intensive Care Unit can cause long-term problems and physiological changes at the neuromuscular and respiratory levels in critically ill patients. Early physiotherapy in these patients is safe and feasible to avoid or reduce the adverse musculoskeletal and respiratory effects of the stay in this hospital unit.

Objective. To identify the strengths and barriers of Physiotherapy in an Intensive Care Unit, according to the vision of different Health Science professionals.

Method. Qualitative observational study using individual interviews and focus groups. 18 people (6 doctors, 6 nurses and 6 physiotherapists) will be included in the study. The 18 health professionals will participate in personal interviews and focus groups (3 focus groups with 6 participants each). Participants will be recruited from the Intensive Care Unit of the Hospital Universitario Central de Asturias. Data will be analysed using the thematic analysis approach according to Braun and Clarke's method. We will use face-to-face interviews and focus groups to collect data and analyse them through thematic analysis. Purposive sampling will be used to recruit our participants. We will continue to recruit participants, if necessary, until saturation of data from the thematic analysis is reached.

Expected outcomes. To assess the knowledge, perceptions and expectations of the healthcare staff in the Intensive Care Unit regarding Physiotherapy in the management of patients admitted to this Unit. To identify the strengths of Physiotherapy in the management of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Professionals from the Intensive Care Unit of the Hospital Universitario Central de Asturias.
* With clinical experience of at least 2 years.
* Currently working or having worked in coordination with physiotherapists in the Intensive Care Unit.

Exclusion Criteria:

* Professionals who are unfamiliar with the usual physiotherapy therapy in an Intensive Care Unit.
* Resident interns in their first year of training.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: To protect the privacy of the healthcare professionals, we will invite the Heads of Service and Section of the Intensive Care Unit to approach potential participants who, based on their personal and clinical experience, may be able to participate in the study. Subsequently, we will schedule a time for personal interviews and focus groups if potential participants are interested in taking part in the study. With the support of the Intensive Care Unit managers, we will be able to recruit healthcare professionals who meet the selection criteria.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2024-05-09 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Assess the knowledge on Physiotherapy in the Intensive Care Unit | Screening visit
  Through open questions focused on the knowledge of physiotherapy in the hospital setting of the Intensive Care Unit: "Are you familiar with the presence of physiotherapists in ICUs?", "Have you previously worked in an ICU that includes physiotherapists?", "Once a patient is admitted to the ICU, when should the physiotherapy intervention start? And when does it actually start?", "What do you think are and should be the functions of physiotherapists in the ICU?", "What do you think are and should be the functions of physiotherapists in the ICU?
Assess the benefits on Physiotherapy in the Intensive Care Unit | Screening visit
  Through open questions focused on the benefits of physiotherapy in the hospital environment of the Intensive Care Unit: "What do you think are the benefits for patients of having physiotherapists in the ICU?", "From the point of view of the work of the physiotherapist, what benefits do you consider most important for the patients admitted to the ICU?", "From the point of view of the work of the physiotherapist, what benefits do you consider most important to facilitate multidisciplinary work in the ICU?"
Assess the collaboration between healthcare professionals in the Intensive Care Unit | Screening visit
  Through open questions focused on the collaboration between healthcare professionals in the Intensive Care Unit: "Have you experienced any challenges in the collaboration between the professionals involved in ICU care in relation to physiotherapy?", "How do you think multidisciplinary collaboration between healthcare professionals in the ICU and the physiotherapists working in the ICU could be improved?
Assess the needs and recommendations of Physiotherapy in the Intensive Care Unit. | Screening visit
  Through open questions focused on the needs and recommendations of Physiotherapy in the Intensive Care Unit: "What additional resources or support do you consider necessary to optimise the presence of physiotherapists in the ICU?", "Do you have any specific recommendations to improve the integration of physiotherapists in the care of patients admitted to the ICU?

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oviedo, Oviedo, Principality of Asturias, Spain

IPD SHARING:
Plan to Share IPD: Undecided